CLINICAL TRIAL: NCT01075165
Title: The Efficacy of Spray Silicone in the Alteration of Physical Burn Scar Characteristics: A Double Blinded Randomized Controlled Trial
Brief Title: Efficacy of Spray Silicone in Alteration of Burn Scar
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB closed study due to no enrollment over 4 yrs
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H-09-041
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Burn Scar
Keywords: silicone; burn scar; hypertrophic scar; keloid; scar assessment; abnormal scarring; Burn patients
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silicone Spray (Experimental): Apply spray silicone
  Interventions: Other: silicone spray
- Saline Spray (Placebo Comparator): Apply Saline Spray
  Interventions: Other: saline spray

INTERVENTIONS:
Other: silicone spray — application of silicone spray to predefined area qd 12 weeks
  Arms: Silicone Spray
Other: saline spray — application of saline spray to predefined area qd 12 weeks
  Arms: Saline Spray

SUMMARY:
In a burn population, conduct a prospective, double-blinded, randomized, controlled clinical trial to determine the ability of spray silicone to alter the physical characteristics of burn scar compared to a placebo.

DETAILED DESCRIPTION:
At study enrollment, the patient's scar will be evaluated using the vascularity category of the Vancouver Scar Scale. The vascularity rating is a four item likert scale that rates the scar as normal (0), pink (1), red (2), or purple (3). Scar height will be measured using a diagnostic ultrasound unit with a 20MHz transducer.27 Digital photographs will be taken with a color spectrum scale placed next to the scar. Laser Doppler imaging (LDI) will be used to assess scar perfusion at the regions of interest to determine whether treatment with silicone spay results in measureable changes in scar perfusion as well as to establish the time course over which these changes may be expected to occur. A spray template will then be created for the patient using thermoplastic material. It will consist of three (3) circles with an area of .785 inches, spaced one inch apart, which will section off the test areas. One of the areas will be treated with the spray silicone, one area will be sprayed with spray saline (to serve as a placebo), the remaining area will not be treated and therefore will serve as the control. The order in which each area is treated will be determined using a randomized block, computerized allocation developed by the study statistician. The spray silicone and spray saline will be applied via containers that conceal the contents and the patients will not be allowed to observe the application of the silicone or saline. Although the patient will be blinded to the test areas that have substances applied to them, there will be no blinding in regard to the control area that receives no treatment. The substances will be applied by trained investigators each weekday for a 12-week period to ensure the method of application is consistent. Both substances will be applied at a distance of 1.5 inches from the surface of the skin for a one second period. Patients will be instructed not to wash the treated area for 24 hours and not to apply pressure garments over the area. The treated areas will be re-evaluated and photographed every two weeks for a 12 week period. The clinician conducting the initial scar evaluation and re-evaluations will be blinded to the scar treatment. Each patient will also complete a scar assessment scale.28 The patient's participation in the study will be concluded 12 weeks after the initial treatment and he/she will be given the option of continued use of the spray silicone, resumption/commencement of pressure garment use or the provision of another appropriate scar management program. Because burn scar can take several months to years to reach the scar maturation phase, the patient will still be a candidate for an alternate scar management program if at the conclusion of this study they see no benefit from the use of spray silicone. If at any time during the 12-week period the clinician determines that the scar is worsening, then the patient will be removed from the study and offered another scar management program.

ELIGIBILITY:
Inclusion Criteria:

1. Military or civilian
2. Between 18-60 years of age
3. Subjects have experienced a deep partial thickness burn injury with a minimal size 2x6 inches in dimension
4. Burn wounds must have healed by secondary intention
5. Available for initial scar evaluation and bi-weekly assessments (30 minutes) and application of silicone and saline every weekday (5 minutes)

Exclusion Criteria:

1. <18 or >60 years
2. Available burn scar size is less then 2x6 inches
3. Burn wounds healed by sheet grafting
4. Unavailable for initial scar evaluation and bi-weekly assessments (30 minutes) and application of silicone and saline every weekday (5 minutes)
5. Pre-existing medical conditions that have the potential to impair healing (i.e. Diabetes, Peripheral Arterial Disease, etc).
6. Pregnant women will be excluded from the study because of the potential for pregnancy hormones to exacerbate the burn scar

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Vascularity rating, scar height, and color of burn scar (spray silicone vs placebo vs untreated) | every 2 weeks for a 12 week period

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - US Army Institute of Surgical Research, Fort Sam Houston, Texas
  - USAISR, Fort Sam Houston, Texas